CLINICAL TRIAL: NCT01449318
Title: Predictors of Postoperative Pain Following Abdominal Hysterectomy
Brief Title: Predictors of Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ANES.MA.13; AUBMC (Other: AUBMC)
Record Dates: First submitted 2011-09-28; First posted 2011-10-10 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2013-09

CONDITIONS: Postoperative Pain
Keywords: Pain; quantitative sensory testing
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients undergoing hysterectomy (No Intervention)
  Interventions: Device: Thermal Sensory Analyzer (Senselab)

INTERVENTIONS:
Device: Thermal Sensory Analyzer (Senselab) — Thermal stimuli will be administered to the ventral surface of the dominant forearm and then to the lower abdomen (surgical site)using the Thermal Sensory Analyser. Each thermal testing trial will be separated by approximately 2 min and at a separate site.
  To measure the thermal pain threshold temperature, The thermode will be applied to the ventral surface of the dominant forearm and the temperature will be increased at 1°C/s from 35 to 50°C.
  To measure the Suprathreshold Thermal Pain Intensity and unpleasantness, Stimulus responses for noxious heat stimuli will be performed by applying phasic heat stimuli at 8 different temperatures (35, 43, 44, 45, 46, 47, 48, and 49°C).
  Other Names: Modular Sensory Analyzer, Senselab

SUMMARY:
The purpose of the study is to prove that pain scores generated from painful stimuli applied preoperatively may help identify the inter-individual variability in pain perception.

DETAILED DESCRIPTION:
Psychological factors and experimental pain models such as as electrical, pressure, heat, or cold stimuli have been identified as predictors of pain intensity and opioid consumption postoperatively. This study will investigate, in addition to the factors described above, the ability of pain scores generated from painful stimuli postoperatively in predicting postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing abdominal hysterectomy through a pfannenstiel incision
* American Society of Anesthesiologists (ASA)Class I-III

Exclusion Criteria:

* Patients with a history of psychiatric disease
* Diabetic or alcoholic patients who may have impaired sensation due peripheral neuropathies
* chronic opioid or nonsteroidal antiinflammatory drug use
* chronic pain conditions

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
pain scores from IV insertion | 15 minutes prior to induction

SECONDARY OUTCOMES:
Anxiety | 24 to 48 hours before surgery
Pain from thermal stimuli | 24 to 48 hours before surgery
  Pain from thermal stimuli will be measure at two sites: site of surgery and at the forearm.
Suprathreshold Thermal pain intensity | 24 to 48 hours before surgery
  Suprathreshold Thermal pain intensity will be recorded at two site: site of surgery and forearm
suprathreshold thermal unpleasantness intensity | 24 to 48 hours before surgery
Expectation about pain | 24 to 48 hours before surgery
postoperative pain | within 1-2 hours after arrival to recovery room; and at 12 hours, 24 hours, 36 hours and 48 hours after surgery
  Postoperative pain will be measured upon arrival to the Post Anesthesia Care Unit (PACU)before morphine consumption and after morphine consumption, at rest and at movement.
Morphine consumption | within 1-2 hours after arrival to recovery room; and at 12 hours, 24 hours, 36 hours and 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marie T Aouad, MD, Principal Investigator — American University of Beirut Medical Center
Locations (2):
- Lebanon (2):
  - American Unversity of Beirut Medical Center, Beirut
  - AUBMC, Beirut